CLINICAL TRIAL: NCT03351361
Title: Randomized Phase III Study Testing Nivolumab and Ipilimumab Versus a Carboplatin Based Doublet in First Line Treatment of PS 2 or Elderly (More Than 70 Years Old) Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Nivolumab and Ipilimumab Versus Chimiotherapy in First Line Treatment in PS 2 or Elderly in Advanced NSCLC Patients
Acronym: eNERGY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-002842-60; 35RC16_9734 (Other: CHU Rennes); 08-2015 (Other: GFPC); CA209-449 (Other: BMS)
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Advanced Non Small Cell Lung Cancer
MeSH Terms: interventions — Nivolumab; Ipilimumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: Nivolumab + Ipilimumab
- Chemotherapy (Active Comparator): carboplatin and pemetrexed or carboplatin and paclitaxel
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Nivolumab + Ipilimumab — Nivolumab dosed intravenously over 30 minutes at 240 mg every 2 weeks combined with Ipilimumab dosed intravenously over 30 minutes at 1 mg/kg every 6 weeks until disease progression, unacceptable toxicity, or other reasons specified in the protocol.
  Arms: Nivolumab + Ipilimumab
Drug: Chemotherapy — Doublet of chemotherapy according to standard of care carboplatin (AUC 5) with a dose that will be capped to 700 mg and pemetrexed (500 mg/m²) over 4 to 6 hours every three weeks (restricted to non-squamous histology) or carboplatin (AUC 6) with a dose that will be capped to 700 mg and paclitaxel (90 mg/m²) D1 D8 D15 over 4 to 6 hours every 4 weeks, with a maximum of 4 cycles of carboplatin based doublet, and the possibility to use maintenance with pemetrexed.
  Arms: Chemotherapy

SUMMARY:
Lung cancer is the most common cancer in the world and the leading cause of cancer-related deaths in Western countries. Unfortunately, at the time of diagnosis, the majority of patients already have metastatic disease and a systemic, palliative treatment is the primary therapeutic option.

Guidelines for PS 2 patients or older than 75 years old patients at the time of diagnosis recommend for fit patients a carboplatin doublet chemotherapy.

Nivolumab has proven efficacy in 3rd line squamous cell lung carcinoma and is superior to chemotherapy in 2nd line treatment of squamous and non-squamous lung cancer in term of overall survival.

In 1st line, nivolumab failed to show superiority compared to a platin based doublet in terms of progression free survival and overall survival in tumors ≥ 5% PD-L1 expression. The association Nivolumab plus Ipilimumab showed encouraging results in first line setting in phase 1 study.

The investigators think that with regard to the manageable toxicity of nivolumab in lung cancer population and the possibility to obtain long responses, this association could be a valid option for this population of elderly and/or PS2 patients in term of overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Cytologically or histologically proven NSCLC (adenocarcinoma, squamous cell carcinoma, large-cell carcinoma)
* Stage IV or non-treatable by radiotherapy or surgery stage III (7th classification)
* No previous systemic chemotherapy for lung cancer, except in case of relapse after adjuvant treatment for localized disease with 6 months or more between end of previous chemotherapy and relapse
* Patients less than 70 years old and PS 2 or 70 years older PS 0 to 2
* Judged fit enough to receive a carboplatin based doublet according to ESMO guidelines
* Presence of at least one measurable target lesion (RECIST 1.1 rules) in a non-irradiated region and analysable by CT
* Life expectancy superior at 12 weeks
* Prior radiation therapy is authorized if it involved less than 25% of the total bone marrow volume and finished 14 days before D1 of planned treatment
* Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization/registration WBC superior or equal at at 2000/μL Neutrophils superior or equal at at 1500/μL Platelets superior or equal at at 100 x103/μL Hemoglobin superior at 10.0 g/dL Serum creatinine inferior or equal at 1.5 x ULN or creatinine clearance (CrCl) superior or equal at at 45 mL/min (if using the Cockcroft-Gault formula ) AST/ALT inferior or equal at 3 x ULN Total Bilirubin inferior or equal at 1.5 x ULN (except Patients with Gilbert Syndrome, who can have total bilirubin inferior at 3.0 mg/dL)
* Availability of adequate FFPE tumor-derived material (tumor blocks or slides) from a biopsy, surgery or fine needle aspirate for analysis of PD-L1 testing by IHC

Age and Reproductive Status

• Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception during treatment.

WOCBP should use an adequate method to avoid pregnancy :

* For 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of nivolumab + ipilimumab,
* For 4 weeks after the last dose of carboplatine + pemetrexed,
* For 5 weeks after the last dose of carboplatine + paclitaxel.

  * Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of treatment
  * Women must not be breastfeeding
  * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year during treatment Men will be instructed to adhere to contraception for a period of 31 weeks after the last dose of nivolumab + ipilimumab and with carboplatine +pemetrexed or carboplatine + paclitaxel up to 6 months thereafter.

Exclusion Criteria:

* Patients with other severe concurrent disorders that occurred during the prior six months before enrollment (myocardial infection, severe or unstable angor, coronarian or peripheric arterial bypass operation, NYHA class 3 or 4 congestive heart failure, transient or constituted cerebral ischemic attack, at least grade 2 peripheral neuropathy, psychiatric or neurological disorders preventing the patient from understanding the trial, uncontrolled infections) are not eligible.
* Serious or uncontrolled systemic disease judged as incompatible with the protocol by the investigator
* Another previous or concomitant cancer, except for basocellular cancer of the skin or treated cervical cancer in situ, or appropriately treated localized low-grade prostate cancer (Gleason score inferior at 6), unless the initial tumor was diagnosed and definitively treated more than 5 years previously, with no evidence of relapse.
* Known activating mutation of EGFR (del LREA exon 19, mutation L858R or L861X of exon 21, mutation G719A/S in exon 18) or EML4-ALK or ROS-1 translocation
* Superior at caval syndrome
* Uncontrolled infectious status
* All concurrent radiotherapy
* Concurrent administration of one or several other anti-tumor therapies.
* Psychological, familial, social or geographic difficulties preventing follow-up as defined by the protocol.
* Protected person (adults legally protected (under judicial protection, guardianship or supervision), person deprived of their liberty, pregnant woman, lactating woman and minor),
* Concurrent participation in another clinical trial
* Patients are excluded if they have active brain metastases or leptomeningeal metastases. Patients with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is 4 weeks or more] after treatment is complete and within 28 days prior to the first dose of nivolumab and ipilimumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (superior at 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration.
* Patients should be excluded if they have an active, known or suspected autoimmune disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (superior at 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses superior at 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients should be excluded if they are positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Patients should be excluded if they have a lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Allergies and Adverse Drug Reaction
* History of allergy to study drug components
* Severe spinal hypoplasia and / or hemorrhagic tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of date of death from any cause, whichever came first, assessed up to 3 years maximum

SECONDARY OUTCOMES:
Survival rate | 1 year
Objective response rate | 2 years
  according to RECIST 1.1
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years maximum
Safety rate | 2 years
  Incidence of Treatment-Emergent Adverse Events according to CTCAE version 4.0
Tolerability rate | 2 years
  Incidence of Treatment-Emergent Adverse Events according to CTCAE version 4.0
Quality of life score | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years maximum
  according to EQ-5D questionnaire
Quality of life score | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years maximum
  according to EORTC QLQ-ELD14 questionnaire
PD-L1 | 2 years
  testing by immunochemistry
Geriatric evaluation | inclusion and 2 months
  according to geriatric mini data set

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Léna, Principal Investigator — CHU Rennes
Locations (30):
- France (30):
  - CH du Pays d'Aix, Aix-en-Provence
  - CHU d'Angers, Angers
  - CH de Beauvais, Beauvais
  - CHU de Brest, Brest
  - Centre Francois Baclesse, Caen
  - CH René Dubos, Cergy-Pontoise
  - CH de Charleville-Mézières, Charleville-Mézières
  - HIA Percy, Clamart
  - CH Intercommunal, Créteil
  - CH Intercommunal des Alpes du Sud, Gap
  - CH Départemental Vendée, La Roche-sur-Yon
  - CH de Versailles, Le Chesnay
  - CH Robert Boulin, Libourne
  - CHU de Limoges, Limoges
  - CH de Bretagne Sud, Lorient
  - Centre Léon Bérard, Lyon
  - CH François Quesnay, Mantes-la-Jolie
  - APHM Hôpital Nord, Marseille
  - Hôpital Européen, Marseille
  - Institut Paoli-Calmette, Marseille
  - CH de Meaux, Meaux
  - CH de la Région d'Annecy, Pringy
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CH de Saint-Brieuc, Saint-Brieuc
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - CLCC Paul Strauss, Strasbourg
  - CH Intercommunal Toulon-La Seyne-sur-Mer, Toulon
  - HIA Saint-Anne, Toulon
  - CH de Villefranche sur Saône, Villefranche-sur-Saône

REFERENCES:
- [Derived] Lena H, Greillier L, Cropet C, Bylicki O, Monnet I, Audigier-Valette C, Falchero L, Vergnenegre A, Demontrond P, Geier M, Guisier F, Hominal S, Locher C, Corre R, Chouaid C, Ricordel C; GFPC 08-2015 ENERGY investigators. Nivolumab plus ipilimumab versus carboplatin-based doublet as first-line treatment for patients with advanced non-small-cell lung cancer aged >/=70 years or with an ECOG performance status of 2 (GFPC 08-2015 ENERGY): a randomised, open-label, phase 3 study. Lancet Respir Med. 2025 Feb;13(2):141-152. doi: 10.1016/S2213-2600(24)00264-9. Epub 2024 Oct 29. PMID 39486424
- [Derived] Gijtenbeek RG, de Jong K, Venmans BJ, van Vollenhoven FH, Ten Brinke A, Van der Wekken AJ, van Geffen WH. Best first-line therapy for people with advanced non-small cell lung cancer, performance status 2 without a targetable mutation or with an unknown mutation status. Cochrane Database Syst Rev. 2023 Jul 7;7(7):CD013382. doi: 10.1002/14651858.CD013382.pub2. PMID 37419867

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03351361/Prot_SAP_001.pdf
  • Informed Consent Form (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03351361/ICF_000.pdf